CLINICAL TRIAL: NCT04608162
Title: Long-term Effect of Electromagnetic Field in Treatment of Patients With Osteopenia or Osteoporosis. A Randomized Placebo-controlled Trial.
Brief Title: Long-term Effect of Electromagnetic Field in Treatment of Patients With Osteopenia or Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm Al-Qura Uni
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Osteopenia or Osteoprosis
Keywords: T-scores of ≤ ˗1.5
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): Group one received PEMF and exercise (PEMF+EX)
  Interventions: Other: Pulsed Electromagnetic Field (PEMF); Other: Exercise Program
- Group II (Placebo Comparator): Group two received placebo PEMF and exercise (PPEMF+EX)
  Interventions: Other: Exercise Program; Other: Placebo PEMF
- Group III (Active Comparator): Group three will be treated by PEMF alone (PEMF)
  Interventions: Other: Pulsed Electromagnetic Field (PEMF)

INTERVENTIONS:
Other: Pulsed Electromagnetic Field (PEMF) — PEMF was administered to the whole body using a 1.8×0.6m mat
  Arms: Group I; Group III
Other: Exercise Program — Exercise program to facilitate bone health
  Arms: Group I; Group II
Other: Placebo PEMF — Patients received placebo PEMF
  Arms: Group II

SUMMARY:
Osteoporosis is the most prevalent metabolic bone disease. Although osteoporosis is widely considered to be much more prevalent in women approximately 39% of new osteoporotic fractures estimated to have occurred worldwide in 2000 were in men. A number of studies investigate the effect of physical therapy modalities in treatment of osteoporosis. The use of pulsed electromagnetic field (PEMF) represents an attractive alternative for osteoporosis.

Previous studies suggested that pulsed electromagnetic field could be beneficial for increase bone mineral density in osteoporotic patients, but there is a lack of knowledge about the long term effect on several parameters.

DETAILED DESCRIPTION:
Objectives: This randomized controlled study aims to investigate the long term effect of pulsed electromagnetic field (PEMF) on bone mineral density (BMD) and bone markers; also to be used as treatment intervention of osteopenia or osteoporosis through studying the effect of low intensity, low frequency, single pulsed electromagnetic fields. Methods: One hundred and twenty male patients with osteopenia or osteoporosis will participate in this study, their age ranges between 30-60 years. They have BMD T-scores ≤ - 1.5. All patients will be randomized into one of three groups. Group one received PEMF and exercise (PEMF+EX), group two received placebo PEMF and exercise (PPEMF+EX) and group three will be treated by PEMF alone (PEMF). The exercise training program will include treadmill and aerobic exercises for hip and upper limb will be performed for 50 minutes.PEMF was administered to the whole body for PEMF groups using a 1.8×0.6m mat 30 minutes/day, 3 times/week for 3 months. Dual-energy X-ray absorptiometry (DEXA) will assess Bone mineral density BMD (g/cm2), bone mineral content (BMC), T-Score and Z-Score at the lumbar spine, proximal femur and forearm region, bone markers (25-hydroxy Vit D , Total, undercarboxylated Ostocalcin, Parathyroid Hormone, Total and Ionized calcium and Alkaline Phosphatase (ALP), also will be measured. The assessment will be done at baseline, after treatment (12 weeks) and after 6 months as follow up. The data will be analyzed using repeated measures Analysis of variance (ANOVA) for comparison between pre-treatment and post treatment measurement intervals. One-way ANOVA is used to compare between each treatment interval in treatment groups at pre-test and post treatment measurement intervals. The level of significance is set at 0.05 for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a T-scores of ≤ ˗1.5, all patients received the same medical treatment for osteoporosis and the same average blood glucose level, sufficient ability to understand the nature and potential risks of the study.

Exclusion Criteria:

* Diabetes mellitus, ischemic heart disease, arrhythmia, uncontrolled thyroid disease, cardiac pacemaker, tuberculosis, neuropsychiatric disorders (dementia, cerebrovascular disease, alcohol abuse, severe depression, panic disorder, bipolar disorder, or psychosis), and malignancy.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline Bone Mineral Density at 3 months | Baseline and 3 months, and 6 months post-intervention
  Bone Mineral Density will assessed by the DEXA in the lumbar spine, proximal femur and forearm region in g/cm2.
Change from baseline Vitamin D levels at 3 months | Baseline and 3 months, and 6 months post-intervention
  Vitamin D test is the most accurate way to measure how much vitamin D is in the body. Vitamin D in serum will measured as a standard procedure at the Department of Clinical Chemistry.
Change from baseline Alkaline Phosphatase at 3 months | Baseline and 3 months, and 6 months post-intervention
  Alkaline Phosphatase will be estimated colorimetric end point and kinetic using fully automated analyzer Advia Centaur, according to enclosed pamphlet.

SECONDARY OUTCOMES:
Change from baseline Osteocalcin at 3 months | Baseline and 3 months, and 6 months post-intervention
  Ostocalcin is a predictive marker for osteoprosis and bone fracture. Serum Osteocalcin will measured in serum samples using an ELISA Kits.
Change from baseline Parathyroid Hormone at 3 months | Baseline and 3 months, and 6 months post-intervention
  Parathyroid hormones (PTH) will measurement chemiluminescence immunoassays [QuiCkIntraOperativeTM intact PTH. The assay will performed on the Immuno- automated analyzer (DPC) at the Department of Clinical Chemistry at Um ALQURA University, Faculty of Applied Medical Science. The Roche intact-PTH test will be assayed on an Elecsys-1010 immunoassay analyzer (Roche Diagnostics) with its "Stat-function.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M El-Shamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Al Noor Specialized Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No